CLINICAL TRIAL: NCT02144337
Title: The Feasibility of a Physical Activity Intervention for Children With Type 1 Diabetes Mellitus: Steps To Active Kids (STAK)
Brief Title: Physical Activity in Children With Type 1 Diabetes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 14005
Record Dates: First submitted 2014-01-16; First posted 2014-05-22 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Type 1 Diabetes Mellitus; Physical Activity
Keywords: Physical activity; Type 1 Diabetes Mellitus; Children; Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Steps To Active Kids (STAK) programme (6 weeks) includes: StreetDance DVD designed to be completed at home (4 weeks in total). A dance routine is taught over 4 weeks with new elements introduced each day. Activity diary aims to encourage children to record daily activities in a logbook and to educate children about physical activity. Step counter: Children are given a pedometer and encouraged to record steps in the activity diary and to set personal goals to increase their steps. Weekly group activity sessions for 4 - 6 weeks. Involve a circuit of activity stations varying in intensity. The group sessions are designed to be fun and non-competitive. Children can record their scores at each station and monitor their own progress.
  Interventions: Behavioral: Steps To Active Kids (STAK) programme
- Control group (No Intervention): Control group. Children in the Control group are asked to continue normal daily activities.

INTERVENTIONS:
Behavioral: Steps To Active Kids (STAK) programme — Intervention described in Arm/Group Description.
  Arms: Intervention group

SUMMARY:
This study aims to test the feasibility of a physical activity intervention called the Steps To Active Kids (STAK) programme in children aged 9 - 11 years with Type 1 Diabetes Mellitus (T1DM).

DETAILED DESCRIPTION:
The STAK programme promotes physical activity in children who have a chronic condition, low levels of physical activity, are overweight or who lack confidence to take part in physical activity. The intervention involves an Activity Diary, circuit training, pedometer step counting, daily physical activity monitoring and goal setting to promote long-term increases in physical activity and its associated health benefits. This randomised single-centre feasibility study will test whether the STAK programme is feasible for children with T1DM, in terms of acceptability, attractiveness and compliance and a qualitative process evaluation will aid the assessment of feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 9 and 11 years
* Have a clinical diagnosis of Type 1 Diabetes Mellitus for at least 3 months
* Be willing and able to comply with the study protocol
* Be physically able to participate in physical activity
* Have a parent/carer who provides informed consent

Exclusion Criteria:

* Be under the age of 9 years and over the age of 11 years
* Have been diagnosed with Type 1 Diabetes Mellitus for less than 3 months
* Have an injury or physical health condition that precludes their participation in physical activity
* Have a psychiatric disorder that interferes with provision of assent, completion of measurements, intervention, or follow-up
* Insufficient proficiency in English to comply with treatment or provide data

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Blake, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals Nhs Trust, Nottingham, United Kingdom

REFERENCES:
- [Derived] Quirk H, Glazebrook C, Blake H. A physical activity intervention for children with type 1 diabetes- steps to active kids with diabetes (STAK-D): a feasibility study. BMC Pediatr. 2018 Feb 7;18(1):37. doi: 10.1186/s12887-018-1036-8. PMID 29415687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment through clinic (single-centre). Postal invitation to all children meeting eligibility criteria.
Pre-assignment Details: Expression of interest request. Consent (parental) and assent (child) received from those who expressed an interest and agreed to participate.
Groups:
- Intervention Group: 6 week Steps To Active Kids (STAK) programme includes: StreetDance DVD designed to be completed at home (4 weeks in total). A dance routine is taught over 4 weeks with new elements introduced each day. Activity diary aims to encourage children to record daily activities in a logbook and to educate children about physical activity. Step counter: Children are given a pedometer and encouraged to record steps in the activity diary and to set personal goals to increase their steps. Weekly group activity sessions for 4 - 6 weeks. Involve a circuit of activity stations varying in intensity. The group sessions are designed to be fun and non-competitive. Children can record their scores at each station and monitor their own progress.
Period: Baseline 0 Months
Arm/Group | Intervention Group | Control Group
Started | 8 | 5
Completed | 8 | 5
Not Completed | 0 | 0
Period: T2 Follow-up (Post-intervention)
Arm/Group | Intervention Group | Control Group
Started | 8 | 5
Completed | 4 | 4
Not Completed | 4 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: T3 Follow-up (3 Month Post-intervention)
Arm/Group | Intervention Group | Control Group
Started | 8 (Number not the same as number who completed previous period due to absence/loss of data at T2) | 5 (Number not the same as number who completed previous period due to absence/loss of data at T2)
Completed | 5 | 5
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants were included in the analysis.
Groups:
- Steps To Active Kids (STAK) Programme: 6 week Steps To Active Kids (STAK) physical activity programme (combined supervised and home-based physical activity).
  Steps To Active Kids (STAK) Programme: 6 week programme of combined supervised and home-based (non-supervised) physical activity.
- Normal Daily Activity: Treatment as usual: children asked to continue normal daily activity as usual.
- Total: Total of all reporting groups
Arm/Group | Steps To Active Kids (STAK) Programme | Normal Daily Activity | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (0.8) | 10.0 (1) | 10.1 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 0 | 6
  Male | 2 | 5 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  White British | 6 | 5 | 11
  Black African | 1 | 0 | 1
  Mixed race | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (calculated from height (cm) and weight (kg) measures from clinic records)
  kg/m^2 | 19.5 (3.8) | 20.5 (3.4) | 19.9 (3.5)
Years diagnosed [Mean (Standard Deviation); unit: years] | 5.1 (3.1) | 2.9 (2.3) | 4.3 (2.9)
Self-reported physical activity [Mean (Standard Deviation); unit: units on a scale] — Children rate a range of activities on a three-point scale representing how much of that activity they did (none, a little, a lot) at three time points in the previous 24 hours; today before school (22 items), yesterday after school (22 items), and yesterday during school (11 items). Scores are summed to form a total score for physical activities (possible range 41-123). Higher values represent higher physical activity (i.e., better outcome).
  units on a scale | 56.8 (9.1) | 49.8 (5.7) | 54.16 (8.5)
CSAPPA total [Mean (Standard Deviation); unit: units on a scale] — CSAPPA = Children's Self-Perceptions of Adequacy in and Predilection for Physical Activity The CSAPPA scale measures generalised self-efficacy and attitudes towards participation in physical activity. The 19-item CSAPPA scale measures children's perceived adequacy, predilection and enjoyment towards physical activity. Each item is scored from 1 to 4 and total CSAPPA scores range between 19 - 76 with higher scores indicative of greater self-efficacy (i.e., better outcome).
  Total score calculated as the sum of all sub-scales (CSAPPA adequacy + CSAPPA predilection + CSAPPA enjoyment)
  units on a scale | 61.7 (5.7) | 59.3 (9.9) | 60.8 (7.1)
CSAPPA Adequacy [Mean (Standard Deviation); unit: units on a scale] — Perceived adequacy (7 items) refers to the perception of one's ability to achieve some acceptable standard of success, that standard being influenced by the self, parents, peers, teachers and society's expectations. Range of scores 7 - 28, with higher scores indicating higher perceived adequacy (i.e., better outcome).
  units on a scale | 22.4 (1.8) | 20.0 (4.5) | 21.5 (3.1)
CSAPPA Predilection [Mean (Standard Deviation); unit: units on a scale] — Predilection (9 items) refers to the preference for being active over being sedentary when given the choice. Range of scores 9 - 36 with higher scores indicating higher predilection towards physical activity (i.e., better outcome).
  units on a scale | 28.7 (4.0) | 29.0 (5.0) | 28.8 (4.1)
CSAPPA Enjoyment [Mean (Standard Deviation); unit: units on a scale] — Enjoyment (3 items) refers to enjoyment of Physical Education (P.E.) class. Range of scores 2 - 12 with higher scores indicating greater enjoyment of P.E (i.e., better outcome).
  units on a scale | 10.6 (1.7) | 10.3 (1.5) | 10.5 (1.6)
PHFS total [Mean (Standard Deviation); unit: units on a scale] — PHFS = Parents' Hypoglycaemia Fear Survey The 26-item PHFS measured parents' fear of hypoglycaemia and the negative consequences of these episodes, as well as behaviours used to avoid hypoglycaemia and its negative consequences. The measure comprises a behaviour subscale and a worry subscale.
  Total score calculated as the sum of both sub-scales (PHFS Behaviour + PHFS Worry).
  Scores range from 0-104. Higher score indicates greater fear of hypoglycaemia (i.e., worse outcome).
  units on a scale | 42.8 (17.6) | 37.4 (11.5) | 42.7 (13.3)
PHFS Behaviour [Mean (Standard Deviation); unit: units on a scale] — 11 items on the PHFS-behaviour subscale assess the behaviours that parents may engage in as a result of fear of hypoglycaemia (e.g., 'avoid having my child being alone when his/her sugar is likely to be low'). Items refer to diabetes management behaviours parents may perform to reduce the chance of hypoglycaemia, the tendency to keep blood glucose levels high to avoid hypoglycaemia and behaviours aimed at avoiding the negative consequences of hypoglycaemia.
  Scores range from 0-44. Higher score indicates more hypoglycaemia avoidance behaviours (i.e., worse outcome).
  units on a scale | 21.9 (7.5) | 20.2 (2.6) | 21.8 (4.4)
PHFS Worry [Mean (Standard Deviation); unit: units on a scale] — 15 items on the PHFS-worry subscale address specific worries that parents may have in relation to various aspects of hypoglycaemia (e.g., 'child not having food, fruit or juice with him/her'). Items on the worry subscale assess worry about hypoglycaemia occurring when the child is alone or when there is no food or drink available, worry about the child having an accident or physical injury, and worry about the child being unable to function normally. Scores on the worry subscale range from 0-60. Higher score indicates greater worry (i.e., worse outcome).
  units on a scale | 21.2 (14.1) | 17.2 (9.8) | 20.8 (12.2)
HbA1c (mmol/mol) [Mean (Standard Deviation); unit: mmol/mol] — Glycaemic control measured in mmol/mol. UK recommended level for good diabetes control is currently <58mmol/mol for children.
  Higher score indicates worse outcome. Lower score (<58mmol/mol) indicates better outcome.
  mmol/mol | 57.1 (10.2) | 55.4 (11.8) | 56.5 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Response Rate
Description: Number of participants completing outcome measures at T2
Time Frame: Response rate at T2
Measure: Number; unit: number of participants
Groups:
- Intervention Group: Steps To Active Kids (STAK) programme
- Control Group: No intervention
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 8 | 5
number of participants | 4 | 4

2. Primary Outcome: Feasibility: Response Rate
Description: Number of participants completing outcome measures at T3
Time Frame: Response rate at T3
Measure: Number; unit: Number of participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 8 | 5
Number of participants | 5 | 5

3. Primary Outcome: Feasibility: Rate of Adherence to the Intervention
Description: Attendance at physical activity sessions and completion of activity diary Intervention group only as the Control group were not exposed to any intervention.
Time Frame: Participants were monitored for the duration of the STAK programme (6 weeks)
Measure: Number; unit: percentage of the intervention group
Arm/Group | Intervention Group
Number analyzed (Participants) | 8
percentage of the intervention group | 75

4. Secondary Outcome: Change in Children's Self-efficacy Using CSAPPA Scale (Children's Self-Perceptions of Adequacy in and Predilection for Physical Activity)
Time Frame: 0 months (baseline) and 6 months (follow-up)
Reporting Status: Not Posted

5. Secondary Outcome: Change in Children's Level of Physical Activity (Measured Subjectively Via Self-report Questionnaire)
Time Frame: 0 months (baseline) and 6 months (follow-up)
Reporting Status: Not Posted

6. Secondary Outcome: Change in Clinical Outcome Measures (Hba1c, Height, Weight)
Description: Data collected as routine clinic procedure and will be used to assess changes in HbA1c and BMI from baseline to follow-up.
Time Frame: 0 months (baseline) and 6 months (follow-up)
Reporting Status: Not Posted

7. Secondary Outcome: Change in Parental Hypoglycaemia Fear Using the Hypoglycaemia Fear Survey (HFS-Parent)
Time Frame: 0 months (baseline) and 6 months (follow-up)
Reporting Status: Not Posted

8. Primary Outcome: Feasibility: Number of Participants With Adverse Events
Description: Number of participants experiencing and/or reporting adverse events.
Time Frame: Participants were followed from baseline to research completion
Measure: Number; unit: number of participants
Groups:
- Overall Study Group Sample: Intervention and control group combined
Arm/Group | Overall Study Group Sample
Number analyzed (Participants) | 13
number of participants | 0

ADVERSE EVENTS:
Time Frame: Data were collected throughout the course of the research (Baseline to completion).
Arm/Group | Steps To Active Kids (STAK) Programme | Normal Daily Activity
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/8 | 0/5

LIMITATIONS AND CAVEATS:
Analysis and interpretation of secondary outcomes ongoing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes